CLINICAL TRIAL: NCT07323550
Title: Comparing Single and Dual Task Effects in Children With Autism Spectrum Disorder and Typically Developing Children
Brief Title: Single-Dual Task Performance in Children With Autism Spectrum Disorder and Typically Developing Children
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gamze Demircioğlu, Ass.prof., Atlas University
Other Study IDs: 2024-ATLAS-MSEHF-003
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autism; Dual Task
MeSH Terms: conditions — Autistic Disorder | interventions — Single Person

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: The diagnosis of Autism Spectrum Disorder was made by child and adolescent psychiatrists in accordance with the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) diagnostic criteria.
  Interventions: Other: Single- and Dual-Task Condition Assessment
- Typically developing child: A control group consisting of children with normal development, matched to the OSB group in terms of age and gender variables, was included.
  Interventions: Other: Single- and Dual-Task Condition Assessment

INTERVENTIONS:
Other: Single- and Dual-Task Condition Assessment — Participants will perform motor tasks under single-task and dual-task conditions. In the dual-task condition, a concurrent cognitive task will be added to the motor task to increase cognitive load. Performance during these conditions will be assessed to examine the effects of cognitive load on motor performance and postural control. No therapeutic intervention, medication, or device is applied.

SUMMARY:
This study aims to compare the effects of single-task and dual-task conditions on motor performance and postural control in children with Autism Spectrum Disorder (ASD) and typically developing children. Participants' performance under single-task and dual-task conditions involving cognitive load will be evaluated to examine how cognitive demands affect physical task performance in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD) Group:
* Aged between 5 and 16 years
* Diagnosed with mild to moderate Autism Spectrum Disorder based on Childhood Autism Rating Scale (CARS) scores
* Ability to understand basic visual, auditory, and verbal instructions
* Sufficient cognitive capacity to follow dual-task instructions

Typically Developing Control Group:

* Age- and sex-matched with the ASD group
* No history of neurological, psychiatric, sensory, orthopedic, or developmental disorders
* No acute or chronic medical conditions
* No pain complaints during assessment
* Written informed consent obtained from a legal guardian

Exclusion Criteria:

Both Groups:

* History of neurological disorders, epilepsy, or seizures
* Orthopedic or musculoskeletal conditions affecting balance
* Visual or hearing impairments (except corrected vision or hearing with glasses or hearing aids)
* Use of assistive devices for walking or balance
* Use of medications affecting balance or motor performance
* Presence of comorbid psychiatric disorders
* Inability to cooperate adequately during assessment
* Absence from more than two consecutive assessment sessions
* Participation in another intervention program during the study period

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of children aged 5 to 16 years, including children diagnosed with mild to moderate Autism Spectrum Disorder and age- and sex-matched typically developing children. All participants are able to follow basic instructions and complete single-task and dual-task motor assessments. Written informed consent is obtained from the legal guardians of all participants prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
Postural control performance | Day 3
  Postural control will be assessed using the Nintendo Wii Balance Board under both single-task and dual-task conditions. The mean value of center of pressure sway in the medio-lateral and anterior-posterior directions will be calculated during a 30-second quiet standing task with eyes open. Values will be expressed in millimeters (mm).

SECONDARY OUTCOMES:
Walking Performance | Day 3
  Gait performance will be assessed under single-task and dual-task conditions using a sensor-based mobile gait analysis application. The mean walking speed will be calculated during a 6-meter walking task performed at a self-selected comfortable pace. Walking speed values will be expressed in meters per second (m/s).
Motor Performance | Day 3
  Motor performance will be assessed under single-task and dual-task conditions using the Sit-to-Stand App. During a 30-second sit-to-stand test, the mean vertical power will be calculated based on average vertical velocity normalized to body weight. Mean power values will be expressed in watts (W) and used as an indicator of lower extremity muscle performance.
Childhood Autism Rating Scale | Day 1
  The Childhood Autism Rating Scale (CARS) was used to assess autism spectrum disorder and rate its severity. The CASR is an observation-based assessment tool developed by Schopler, Reichler, and Renner in 1980.The scale consists of 15 items and covers behavioral areas such as social relationships, imitation, emotional responses, physical movements, adaptation, visual and auditory responses, olfactory responses, language communication, and intelligence . In the scoring of the test, 15-29 points indicate no signs of autism, 30-37 points indicate mild to moderate levels, and 38-60 points indicate severe levels of autistic traits .

CONTACTS AND LOCATIONS:
Locations (1):
- Moren Language, Speech, and Development Center, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No